CLINICAL TRIAL: NCT04742699
Title: An Open-label, Multicenter Study to Evaluate the Efficacy and Safety of Transitioning to Lemborexant in Japanese Subjects With Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kurume University (Other)
Collaborators: Eisai Inc. (Industry); Mebix Inc (Industry)
Responsible Party: Principal Investigator, Motohiro Ozone, Professor, Kurume University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2006-M081-401
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — lemborexant; leukocyte endogenous mediator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Z-Drug-mono cohort (Experimental): Patients being treated with Z-drug monotherapy at registration
  Interventions: Drug: Lemborexant (LEM) 5 mg (Z-Drug-mono cohort)
- SUV-mono cohort (Experimental): Patients being treated with SUV monotherapy at registration
  Interventions: Drug: Lemborexant (LEM) 5 mg (SUV-mono cohort)
- SUV-combination cohort (Experimental): Patients being treated with SUV and BZRA combination therapy at registration
  Interventions: Drug: Lemborexant (LEM) 5 mg (SUV-combination cohort)
- RMT-combination cohort (Experimental): Patients being treated with RMT and BZRA combination therapy at registration
  Interventions: Drug: Lemborexant (LEM) 5 mg (RMT-combination cohort)

INTERVENTIONS:
Drug: Lemborexant (LEM) 5 mg (Z-Drug-mono cohort) — 1. Pretreatment phase: Continue pre-registration treatment (Z-drug monotherapy) without LEM.
  2. First treatment phase: Administer LEM 5 mg/day as a substitute for Z-Drug. Increasing LEM dose to 10 mg/day is allowed.
  3. Maintenance phase: Succeed the treatment from the first treatment phase. Changing LEM dose is allowed. Rescue administration of Z-drug or RMT is allowed under a defined condition.
  Arms: Z-Drug-mono cohort
Drug: Lemborexant (LEM) 5 mg (SUV-mono cohort) — 1. Pretreatment phase: Continue pre-registration treatment (SUV monotherapy) without LEM.
  2. First treatment phase: Administer LEM 5 mg/day as a substitute for SUV. Increasing to LEM dose to 10 mg/day is allowed.
  3. Maintenance phase: Succeed the treatment of the first treatment phase. Changing LEM dose is allowed.
  Arms: SUV-mono cohort
Drug: Lemborexant (LEM) 5 mg (SUV-combination cohort) — 1. Pretreatment phase: Continue pre-registration treatment (SUV and BZRA combination therapy) without LEM.
  2. First treatment phase: Administer LEM 5 mg/day as a substitute for SUV and continue BZRA. Increasing to LEM dose to 10 mg/day is allowed.
  3. Maintenance phase: Succeed the treatment of the first treatment phase. Changing LEM dose is allowed. Decreasing dose or discontinuation of BZRA is allowed. Rescue administration of Z-drug or RMT is allowed under a defined condition.
  Arms: SUV-combination cohort
Drug: Lemborexant (LEM) 5 mg (RMT-combination cohort) — 1. Pretreatment phase: Continue pre-registration treatment (RMT and BZRA combination therapy) without LEM.
  2. First treatment phase: Administer LEM 5 mg/day as a substitute for RMT and continue BZRA. Increasing to LEM dose to 10 mg/day is allowed.
  3. Maintenance phase: Succeed the treatment of the first treatment phase. Changing LEM dose is allowed. Decreasing dose or discontinuation of BZRA is allowed. Rescue administration of Z-drug or RMT is allowed under a defined condition.
  Arms: RMT-combination cohort

SUMMARY:
This study will be conducted to evaluate whether the approach of direct transitioning to lemborexant (LEM) is supported for insomnia patients who are unsatisfied with current medication.

Transition from Following 4 regimens of interest will be investigated; Z-Drug monotherapy, suvorexant (SUV) monotherapy, SUV and benzodiazepine receptor agonists (BZRA) combination therapy, and ramelteon (RMT) and BZRA combination therapy. Patients with insomnia who have been treated with one of the regimens but do not have treatment satisfaction will be enrolled.

As a comprehensive indicator of patient satisfaction including treatment efficacy and safety, the proportion of patients with successful transitioning will be evaluated at 2 weeks after transitioning; thus important initial response after transitioning will be evaluated as a primary endpoint. In addition, as a secondary purpose, the treatment continuation, efficacy and tolerability, and the treatment impression for insomnia (Patient Global Impression of Insomnia) for 14 weeks after transitioning will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have voluntarily provided a written informed consent to participate in the study
2. Subjects with insomnia aged 20 years or older at the time of informed consent
3. Subjects who are dissatisfied with the efficacy or tolerability of prior medications and wish to transition from them. For example;

   * Subjects who are treated with Z-Drug monotherapy or a combination of BZRA and RMT, and have particularly difficulties with sleep maintenance
   * Subjects who are treated with SUV monotherapy or a combination of BZRA and SUV, and have particularly difficulties with sleep onset
   * Subjects who are treated with a combination therapy of BZRA and SUV or BZRA and RMT, and wish to reduce or discontinue BZRA
4. Subjects with frequent use (i.e. at least 5 nights a week) of Z-drug monotherapy, SUV monotherapy, combination therapy with BZRA and SUV, or combination therapy with BZRA and RMT in the month before the start of the pretreatment phase.
5. Subjects who meet the criteria for insomnia disorder in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) as follows

   * Despite an adequate opportunity for sleep, subjects have night sleep-related complaints accompanied by at least 1 of the following symptoms: difficulty in falling asleep, difficulty in staying asleep, and waking up early
   * The difficulty in sleeping occurs at least 3 nights a week
   * The difficulty in sleeping persists for at least 3 months
   * The difficulty in sleeping causes daytime dysfunction
6. Subjects who can secure at least 7 hours for sleep
7. Subjects who have a documented use of a prior medication(s) for the treatment of insomnia at least 5 nights in the last 2 weeks of the pretreatment phase
8. Subjects who are able to comply with the requirements specified in the study protocol

Exclusion Criteria:

1. Female who are breastfeeding or pregnant at pretreatment phase. If pregnancy cannot be completely denied by interview, a serum beta-hCG test will be performed.
2. Females of childbearing potential who did not use a highly effective method of contraception, which includes:

   * total abstinence (if it is their preferred and usual lifestyle)
   * use of condom
   * an intrauterine device (IUD)
   * a contraceptive implant
   * an oral or an injective contraceptive
   * have a vasectomized partner with confirmed azoospermia; The following methods are not considered as contraception: periodic abstinence such as calendar method, ovulation method, symptothermal method, basal body temperature method, and withdrawal method.
   * Do not agree to use a highly effective method of contraception (as described above)
3. Subjects with moderate or severe obstructive sleep apnea (OSA).
4. Subjects with any symptoms and/or disease that may affect the safety or the endpoints of the study in the opinion of the investigator (see the examples below)

   * Cardiac disorder [including subjects with repeated QT interval prolongation*1 in previous ECG tests. For subjects whose QT interval abnormality cannot be ruled out by interview, ECG tests should be performed by baseline (Visit 2) to confirm the normality of corrected QT (QTc) interval].

     *1: QT interval corrected by Fridericia's formulas (QTcF) exceeds 450 ms
   * Respiratory disorder other than mild OSA
   * Digestive disease
   * Kidney disease [including renal dysfunction]
   * Neurological disorders [including intellectual incapacity or cognitive decline with disorientation to the person, place, time or situation]
   * Mental disorders
   * Chronic pain [pain disorders]
   * Carcinoma within 5 years [excluding appropriately treated basal cell carcinoma]
5. Subjects who currently have certain sleep disorders other than insomnia such as periodic limb movement disorder, restless legs syndrome, and circadian rhythm sleep disorder. Subjects diagnosed with mild OSA are not excluded from the study
6. Subjects who currently have a habit of napping for a long period of time 3 or more times a week in the opinion of the investigator.
7. Subjects who currently have narcolepsy or cataplexy
8. Subjects who are using a prior medication(s) for the treatment of insomnia at doses exceeding the dosage and administration approved in Japan
9. Subjects who are using two or more BZRAs
10. Subjects who are using sedative medication(s)
11. Have used prohibited concomitant drugs within 1 week before the start of the pretreatment phase
12. Have newly started nonpharmacologic treatments for insomnia (eg, cognitive behavioral therapy) within 1 week before the pretreatment phase
13. Subjects who cannot refrain from excessive alcohol consumption during study participation
14. Subjects with a history of hypersensitivity to any of the excipients of LEM
15. Subjects with moderate or severe hepatic impairment (subjects whose AST, ALT, or gamma-GTP is 3 times or more the upper limit of the institutional reference interval)
16. History of antipsychotic drugs use within the past 2 years or attempted suicide, which may affect the safety or the endpoints of the study in the opinion of the investigator
17. Subjects who have previously taken LEM (including subjects who have participated in a clinical trial of LEM)
18. Subjects deemed inappropriate to participate in this study in the opinion of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with successful LEM treatment at the end of the first treatment phase to the patients who started the first treatment phase. | 2 weeks
  The primary endpoint is the proportion of patients with successful LEM treatment at the end of the first treatment phase to the patients who started the first treatment phase. Evaluation is performed for each treatment group.
  Successful LEM treatment at the end of the first treatment phase is primarily defined as follows;
  * Patients who wish to continue LEM treatment at the end of the first treatment phase and actually move on to the maintenance phase
  * Patients who wish to continue LEM treatment at the end of the first treatment phase but do not move to the maintenance phase with a reason not related to the efficacy or safety of LEM treatment (e.g., relocation, clinic transfer, or a burden of site visit expenses)

SECONDARY OUTCOMES:
Proportion of patients who continued LEM treatment and those who continued LEM monotherapy at the end of the first treatment phase and the maintenance phase. | 2 - 14 weeks
Proportion of patients with an itemized positive response on the PGI-I at baseline, the end of the first treatment phase, and the end of the maintenance phase. | 2 - 14 weeks
Proportion of patients with increased LEM dosage at the end of the first treatment phase and at the end of the maintenance phase. | 2 - 14 weeks
Occurrence of adverse events during the first treatment phase and the maintenance phase. | 2 - 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Motohiro Ozone, Principal Investigator — Kurume University
Locations (9):
- Japan (9):
  - YOU ARIYOSHI Sleep Clinic, Kitakyushu, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Hirota Clinic, Kurume, Fukuoka
  - Kurume University Medical Center, Kurume, Fukuoka
  - Kotorii Isahaya Hospital, Isahaya, Nagasaki
  - Ohshima Hospital, Nakatsukuma, Saga-ken
  - Sleep Support Clinic, Shinagawa, Tokyo
  - Sleep & Stress Clinic, Shinagawa, Tokyo
  - Kuwamizu Hospital, Kumamoto

REFERENCES:
- [Derived] Ozone M, Hirota S, Ariyoshi Y, Hayashida K, Ikegami A, Habukawa M, Ohshima H, Harada D, Hiejima H, Kotorii N, Murotani K, Nishi Y, Koebis M, Taninaga T, Uchimura N. Self-reported sleep variables, sleep quality, and quality of life assessment in transition to lemborexant in patients with Insomnia: the multicenter, open-label SOMNUS study. Sleep Med X. 2025 Sep 25;10:100149. doi: 10.1016/j.sleepx.2025.100149. eCollection 2025 Dec 15. PMID 41103818
- [Derived] Ozone M, Hirota S, Ariyoshi Y, Hayashida K, Ikegami A, Habukawa M, Ohshima H, Harada D, Hiejima H, Kotorii N, Murotani K, Taninaga T, Uchimura N. Efficacy and Safety of Transitioning to Lemborexant from Z-drug, Suvorexant, and Ramelteon in Japanese Insomnia Patients: An Open-label, Multicenter Study. Adv Ther. 2024 Apr;41(4):1728-1745. doi: 10.1007/s12325-024-02811-2. Epub 2024 Mar 9. PMID 38460107